CLINICAL TRIAL: NCT01489241
Title: Renewing Health RCT in Central Greece for the Evaluation of Short-term Telehealth Follow up After Hospital Discharge for COPD Exacerbation
Brief Title: Short-term Telehealth Follow up After Hospital Discharge for Chronic Obstructive Pulmonary Disease Exacerbation
Acronym: RHCluster4GR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Health Authority of Sterea & Thessaly (Other Government)
Collaborators: Ministry for Health and Social Solidarity, Greece (Other); Municipality of Trikala, Greece (Other); e-Trikala S.A. (Industry); Cities Net SA (Industry); Institute of Biomedical Research & Technology, Larissa, Greece (Other); Institute of Communications and Computer Systems, Athens, Greece (Other); Alexander Technological Educational Institute, Thessaloniki, Greece (Other); University of Macedonia, Thessaloniki, Greece (Other); University of Thessaly (Other)
Responsible Party: Principal Investigator, Konstantinos Gourgoulianis, Professor, Director of the Pulmonary Department, University Hospital of Larisa, Regional Health Authority of Sterea & Thessaly
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FR2017; EC Grant Agreement 250487 (Other Grant/Funding Number: European Commission CIP/PSP-ICT Grant Agreement 250487)
Record Dates: First submitted 2011-12-06; First posted 2011-12-09 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2015-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Pulmonary Disease, Chronic Obstructive; Telemedicine
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (No Intervention): Patients in the control group receive usual care and visit the outpatient department at 4 and at 12 weeks after discharge when pulse rate, oxygen saturation and spirometry is performed. In the case of clinical deterioration during the study, the patients contact as usual their general practitioner. Usual care of COPD patients consists of regular visits to the specialist or primary care clinics every time a medication change is made or a medical examination is needed
- Telemonitoring (Experimental)
  Interventions: Procedure: Telemonitoring

INTERVENTIONS:
Procedure: Telemonitoring — Within 24 hours after patient's discharge, the telemedicine equipment is installed at the patient's home and patients are trained in the use of the equipment. Patients are followed by a dedicated telehealth centre. Patients at home are asked to fill out each morning the CAT questionnaire and to record extra use of COPD relief medications. Patients in stable conditions perform telespirometry and teleoximetry at 4 and 12 weeks. When a clinical worsening is detected (increase in CAT score by 5 points or higher on two consecutive days) the patient is contacted and asked to perform ad hoc telespirometry and teleoximetry and to send the data to the telehealth centre.
  Arms: Telemonitoring

SUMMARY:
The purpose of this study is to evaluate whether the introduction of a short-term telemonitoring program for chronic obstructive pulmonary disease (COPD) patients discharged from the hospital after disease exacerbation produces benefits in terms of a reduction in hospital readmissions and health related quality of life. In addition the trials evaluate the economical and organisational impact of the services and examine their acceptability by patients and health professionals.

DETAILED DESCRIPTION:
The purpose of this study is to the evaluate the use of a close phone-based tele-monitoring platform will reflected by less hospital re-admissions, will change their generic and disease specific quality of life compared with usual care. Following this; it is also hypothesized that this will also lead to less patients' deaths. In addition the patients' satisfaction using the telemedicine service will be studied. A Cost-Effective Analysis will evaluate the tele-health service compared with the usual care from the health and social perspective.

ELIGIBILITY:
Inclusion Criteria:

* Exacerbation of COPD according to the GOLD guidelines
* Age > 40 years
* Capability to use the devices provided
* Willing to participate

Exclusion Criteria:

included in previous COPD monitoring study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Number of hospital readmissions | 3 months period
  Number of hospital readmissions after the hospital discharged of the patient after a COPD exacerbation

SECONDARY OUTCOMES:
Health related quality of life of the patients as measured by the SF-36 version 2 questionnaire | 3 months - at the entry point of the intervention and the end.
  Health related quality of life of the patients as measured by the SF-36 version 2 questionnaire
Hospital anxiety and depression scale HADS | 3 months - at the entry point of the intervention and the end.
  Hospital anxiety and depression scale HADS
Health status, measured with the St. George's Respiratory Questionnaire SGRQ | 3 months - at the entry point of the intervention and the end.
  Health status, measured with the St. George's Respiratory Questionnaire SGRQ
Lung condition as measured by FEV1 | 1 month after the hospital discharge.
  Lung condition as measured by FEV1
Mortality | 3 months period
  Mortality
Patients' Acceptance-Satisfaction measured by the WSD Questionnaire | at the 3rd month of the tele-monitoring
  Patients' Acceptance-Satisfaction of telemonitoring measured by the Whole System Demonstrators Questionnaire , for the intervention arm (telemonitoring)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Gourgoulianis, MD, PhD, Principal Investigator — Pulmonary Department - University Hospital of Larisa
Locations (1):
- Pulmonary Department - Regional University Hospital of Larisa, Larissa, Thessaly, Greece

REFERENCES:
- [Background] Polisena J, Tran K, Cimon K, Hutton B, McGill S, Palmer K, Scott RE. Home telehealth for chronic obstructive pulmonary disease: a systematic review and meta-analysis. J Telemed Telecare. 2010;16(3):120-7. doi: 10.1258/jtt.2009.090812. Epub 2010 Mar 2. PMID 20197355
- See also: "The Renewing Health project is partially funded under the ICT Policy Support Programme (ICT PSP) as part of the Competitiveness and Innovation Framework Programme by the European Community" — http://www.renewinghealth.eu/